CLINICAL TRIAL: NCT00998257
Title: Regulatory Post Marketing Surveillance Study on YAZ
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 14785; YA0910KR (Other: company internal); YAZ rPMS (Other: company internal)
Record Dates: First submitted 2009-09-21; First posted 2009-10-20 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Contraception; Premenstrual Syndrome; Acne
Keywords: Contraception; Premenstrual Dysphoric Disorder; PMDD; Acne
MeSH Terms: conditions — Premenstrual Syndrome; Acne Vulgaris; Premenstrual Dysphoric Disorder | interventions — drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: EE20/DRSP (YAZ, BAY86-5300)

INTERVENTIONS:
Drug: EE20/DRSP (YAZ, BAY86-5300) — Patients under daily life treatment with YAZ according to local drug information.

SUMMARY:
The objective of this Post Marketing Surveillance (PMS) is to gain information about safety and efficacy in real practice.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects

  * requesting contraception
  * suggesting PMDD by Physician who are also requesting contraception
  * with acne who are also requesting contraception
* Age: 18 - 50 years
* Women who is prescribed YAZ first, during study period

Exclusion Criteria:

* Women who are contraindicated based on the label of YAZ

  * Presence or a history of venous or arterial thrombotic/ thromboembolic events (e.g. deep venous thrombosis, pulmonary embolism, myocardial infarction) or of a cerebrovascular accident
  * Presence or history of prodromi of a thrombosis (e.g. transient ischaemic attack, angina pectoris)
  * History of migraine with focal neurological symptoms
  * Diabetes mellitus with vascular involvement
  * The presence of a severe or multiple risk factor(s) for venous or arterial thrombosis may also constitute a contraindication
  * Pancreatitis or a history thereof if associated with severe hypertriglyceridemia
  * Presence or history of severe hepatic disease as long as liver function values have not returned to normal
  * Severe renal insufficiency or acute renal failure
  * Presence or history of liver tumours (benign or malignant)
  * Known or suspected sex-steroid influenced malignancies (e.g. of the genital organs or the breasts)
  * Undiagnosed vaginal bleeding
  * Known or suspected pregnancy
  * Hypersensitivity to the active substances or to any of the excipients

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Korean female who need only contraception or contraception and management of PMDD or contraception and treatment of acne.
Sampling Method: Non-Probability Sample
Enrollment: 770 (Actual)
Dates: Start 2009-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Adverse event collection | After taking YAZ for 3 cycles and 6 cycles (1 cycle is 28 days)
Contraception efficacy | After taking YAZ for 3 cycles and 6 cycles (1 cycle is 28 days)
Drug compliance | After taking YAZ for 3 cycles and 6 cycles (1 cycle is 28 days)
Release of Premenstrual Dysphoric Disorder (PMDD) or acne | After taking YAZ for 3 cycles and 6 cycles (1 cycle is 28 days)

SECONDARY OUTCOMES:
Number of patients who used YAZ just for contraception | At initial visit (Day 0)
Number of patients who used YAZ for PMDD + contraception | At initial visit (Day 0)
Number of patients who used YAZ for Acne + contraception | At initial visit (Day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, South Korea